CLINICAL TRIAL: NCT04886674
Title: Bovine Colostrum in Prevention of Necrotizing Enterocolitis and Sepsis in Very Low Birth Weight Neonates: a Prospective Study at Neonatology Unit of Children's Hospital Assiut University
Brief Title: Bovine Colostrum in Prevention of Necrotizing Enterocolitis and Sepsis in Very Low Birth Weight Neonates
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Kamal Ali Abd El Hameed, principle investigator, Assiut University
Other Study IDs: Bovine Colostrum in NEC
Record Dates: First submitted 2021-04-22; First posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: NEC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Remuverol: The neonates will receive the colostrum in a dose of 2 g/dose for the 1000-1500 g stratum and 1.2 g/dose for < 1000 g stratum, four times a day until discharge or death or day 21 of life, whichever is earlier.
  Interventions: Dietary Supplement: bovine colostrum

INTERVENTIONS:
Dietary Supplement: bovine colostrum — The neonates will receive the colostrum in a dose of 2 g/dose for the 1000-1500 g stratum and 1.2 g/dose for < 1000 g stratum, four times a day until discharge or death or day 21 of life, whichever is earlier.
  Other Names: placebo

SUMMARY:
Primary Aim: The aim of this study is to investigate the efficacy of bovine colostrum in prevention of necrotizing enterocolitis (NEC) and sepsis in very low birth weight (VLBW) infants.

Secondary Aim: To improve outcomes of neonatal sepsis and NEC in the pe-terrms and to decrease their hospital stay.

DETAILED DESCRIPTION:
Necrotizing enterocolitis (NEC) primarily occurs in premature and very low birth weight (VLBW) babies, the incidence varying from 5 to 10% in various neonatal intensive care unit (NICUs) .

Many researchers believe that an exaggerated inflammatory response mounted by immature intestinal epithelial cells in response to abnormal intestinal colonization plays a vital role in the pathogenesis of NEC and bacteria belonging to Enterobacteriaceae have often been linked to NEC .

Colonization with commensal bacteria soon after birth is essential for the development of normal intestinal function however, this process is often altered in premature babies in NICUs, leading to colonization with pathogenic bacteria .

Commercially available bovine colostrum has high concentrations of anti-infective factors such as immunoglobulins, lactoferrin, organism-specific antibodies, lactoperoxidase, insulin-like growth factors and transforming growth factors.

These components have substantial homology to their human counterparts . Bovine colostrums has been tried in the treatment of Escherichia coli and Shigella and Rotavirus diarrhea in children, Helicobacter pylori infection in children and E. coli intestinal infection in term and preterm neonates.

No major adverse effects were reported in any of the studies using bovine colostrum in infants and preterm babies .

In an in vitro study, the authors showed that bovine colostrum significantly reduces the adherence of various Enterobacteriaceae species known to be associated with NEC to human intestinal epithelial cells .

A randomized controlled trial has shown that the use of bovine lactoferrin reduced the incidence of neonatal sepsis .

Till date, there are no studies in neonates on the use of bovine colostrum for the prevention of NEC.

ELIGIBILITY:
Inclusion Criteria:

* Babies with birth weight ≤ 1500 g

Exclusion Criteria:

* Babies who have any contraindication for initiating milk feeds; who will fail to achieve adequate feed volume to be able to administer the study drug.
* Those with suspected/ proven gastrointestinal malformations.
* Preexisting sepsis (definite or suspect) or NEC at the time of enrollment.
* Those with a family history of an inborn error metabolism (that precludes exposure to proteins/lactose).

Ages: 1 Day to 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The neonates will receive the colostrum in a dose of 2 g/dose for the 1000-1500 g stratum and 1.2 g/dose for < 1000 g stratum, four times a day until discharge or death or day 21 of life, whichever is earlier.
Sampling Method: Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will be definite NEC | baseline
  Subjects who will be suspected to have NEC (based on clinical features) undergo an abdominal X-ray and stool occult blood assay.

SECONDARY OUTCOMES:
Descriptive statistics will be used for describing baseline variables.Dichotomous outcomes will be compared by Chi square test with continuity correction or Fisher's Exact as applicable. | baseline
  Numerical variables will be compared by Student's t-test or Mann Whitney U-test, depending on distribution.

REFERENCES:
- [Background] Thompson AM, Bizzarro MJ. Necrotizing enterocolitis in newborns: pathogenesis, prevention and management. Drugs. 2008;68(9):1227-38. doi: 10.2165/00003495-200868090-00004. PMID 18547133
- [Background] Grave GD, Nelson SA, Walker WA, Moss RL, Dvorak B, Hamilton FA, Higgins R, Raju TN. New therapies and preventive approaches for necrotizing enterocolitis: report of a research planning workshop. Pediatr Res. 2007 Oct;62(4):510-4. doi: 10.1203/PDR.0b013e318142580a. PMID 17667844
- [Background] Hoy CM, Wood CM, Hawkey PM, Puntis JW. Duodenal microflora in very-low-birth-weight neonates and relation to necrotizing enterocolitis. J Clin Microbiol. 2000 Dec;38(12):4539-47. doi: 10.1128/JCM.38.12.4539-4547.2000. PMID 11101593
- [Background] Peter CS, Feuerhahn M, Bohnhorst B, Schlaud M, Ziesing S, von der Hardt H, Poets CF. Necrotising enterocolitis: is there a relationship to specific pathogens? Eur J Pediatr. 1999 Jan;158(1):67-70. doi: 10.1007/s004310051012. PMID 9950312
- [Background] Hoy C, Millar MR, MacKay P, Godwin PG, Langdale V, Levene MI. Quantitative changes in faecal microflora preceding necrotising enterocolitis in premature neonates. Arch Dis Child. 1990 Oct;65(10 Spec No):1057-9. doi: 10.1136/adc.65.10_spec_no.1057. PMID 2122814